CLINICAL TRIAL: NCT03909698
Title: Antibiotic Dosing in Patients on Intermittent Hemodialysis
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: UGent_ABdosing
Record Dates: First submitted 2019-04-04; First posted 2019-04-10 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2021-08

CONDITIONS: Kidney Failure, Chronic; Antibiotics; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sampling of blood and urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Hemodialysis patients on amoxicillin-clavulanic acid: The antibiotic administration protocol is not changed for this study. From the first administration on, administrations (dosage and duration) are well documented. Blood samples are taken as peak, distribution and trough samples during at least 24 or 48 hours. During the first dialysis session after study start, blood samples are also taken from the arterial and venous blood line simultaneously and at different dialysis time points, to calculate dialyzer extraction ratio. When appropriate, urine is collected during a documented period. During the second dialysis after study start, arterial and venous samples are taken for different dialysis settings, in order to calculate extraction ratios for different settings.
  All blood and urine samples are analyzed for amoxicillin-clavulanic acid.
  Interventions: Other: Blood and urine sampling
- Hemodialysis patients on ceftazidim: The antibiotic administration protocol is not changed for this study. From the first administration on, administrations (dosage and duration) are well documented. Blood samples are taken as peak, distribution and trough samples during at least 24 or 48 hours. During the first dialysis session after study start, blood samples are also taken from the arterial and venous blood line simultaneously and at different dialysis time points, to calculate dialyzer extraction ratio. When appropriate, urine is collected during a documented period. During the second dialysis after study start, arterial and venous samples are taken for different dialysis settings, in order to calculate extraction ratios for different settings.
  All blood and urine samples are analyzed for ceftazidim.
  Interventions: Other: Blood and urine sampling
- Hemodialysis patients on piperacillin-tazobactam: The antibiotic administration protocol is not changed for this study. From the first administration on, administrations (dosage and duration) are well documented. Blood samples are taken as peak, distribution and trough samples during at least 24 or 48 hours. During the first dialysis session after study start, blood samples are also taken from the arterial and venous blood line simultaneously and at different dialysis time points, to calculate dialyzer extraction ratio. When appropriate, urine is collected during a documented period. During the second dialysis after study start, arterial and venous samples are taken for different dialysis settings, in order to calculate extraction ratios for different settings.
  All blood and urine samples are analyzed for piperacillin-tazobactam.
  Interventions: Other: Blood and urine sampling
- Hemodialysis patients on vancomycin: The antibiotic administration protocol is not changed for this study. From the first administration on, administrations (dosage and duration) are well documented. Blood samples are taken as peak, distribution and trough samples during at least 24 or 48 hours. During the first dialysis session after study start, blood samples are also taken from the arterial and venous blood line simultaneously and at different dialysis time points, to calculate dialyzer extraction ratio. When appropriate, urine is collected during a documented period. During the second dialysis after study start, arterial and venous samples are taken for different dialysis settings, in order to calculate extraction ratios for different settings.
  All blood and urine samples are analyzed for vancomycin.
  Interventions: Other: Blood and urine sampling
- Hemodialysis patients on teicoplanin: The antibiotic administration protocol is not changed for this study. From the first administration on, administrations (dosage and duration) are well documented. Blood samples are taken as peak, distribution and trough samples during at least 24 or 48 hours. During the first dialysis session after study start, blood samples are also taken from the arterial and venous blood line simultaneously and at different dialysis time points, to calculate dialyzer extraction ratio. When appropriate, urine is collected during a documented period. During the second dialysis after study start, arterial and venous samples are taken for different dialysis settings, in order to calculate extraction ratios for different settings.
  All blood and urine samples are analyzed for teicoplanin.
  Interventions: Other: Blood and urine sampling

INTERVENTIONS:
Other: Blood and urine sampling — During a period of maximum 6 days blood is sampled at different time points and urine is collected during documented time intervals.

SUMMARY:
The adequacy of the currently used dosing regimen of glycopeptides (vancomycin and teicoplanin) and beta-lactam antibiotics (amoxicillin-clavulanic acid, piperacillin-tazobactam, ceftazidim) in patients with end-stage kidney disease receiving intermittent hemodialysis is studied by evaluating pharmacokinetics-pharmacodynamics (PK-PD) target attainment. A population pharmacokinetic study is performed to assist the selection of the optimal individualized dose for patients undergoing intermittent dialysis, taking into consideration as many relevant variables as possible.

ELIGIBILITY:
Inclusion Criteria:

* patients with end-stage kidney disease, requiring intermittent hemodialysis
* patient receiving antibiotic treatment for documented or presumed infection (vancomycin, teicoplanin, amoxicillin-clavulanic acid, piperacillin-tazobactam, ceftazidim)

Exclusion Criteria:

* pregnant woman
* absence of written informed consent from the patient
* known hypersensitivity or contra-indication to glycopeptides or beta-lactam antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Per antibiotic agent, up to 30 patients are included. The final needed number is anticipated by the numer of smamples per patient and the pharmacokinetic modeling.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Blood concentrations with maximal antimicrobial activity versus current dosing regimens for vancomycin | 9/2016 - 12/2021
  Measured free and total concentration of the glycopeptide vancomycin is compared to predefined pharmacokinetic/pharmacodynamic (PK-PD) targets:
  Area Under the Curve (AUC) from 0-24h in steady-state divided by the Minimum Inhibitory Concentration (MIC) of the suspected pathogen should be >=400 for vancomycin.
Blood concentrations with maximal antimicrobial activity versus current dosing regimens for teicoplanin | 9/2016 - 12/2021
  Measured free and total concentration of the glycopeptide teicoplanin is compared to predefined pharmacokinetic/pharmacodynamic (PK-PD) targets:
  Area Under the Curve (AUC) from 0-24h in steady-state divided by the Minimum Inhibitory Concentration (MIC) of the suspected pathogen should be >=750 for teicoplanin.
Blood concentrations with maximal antimicrobial activity versus current dosing regimens for amoxicillin-clavulanic acid | 9/2016 - 12/2021
  Measured concentration of the beta-lactam amoxicillin-clavulanic acid is compared to predefined pharmacokinetic/pharmacodynamic (PK-PD) targets:
  minimum percentage of time during which the free drug concentration remains above the Minimum Inhibitory Concentration (MIC) of the micro-organism should be 50%.
Blood concentrations with maximal antimicrobial activity versus current dosing regimens for piperacillin-tazobactam | 9/2016 - 12/2021
  Measured concentration of the beta-lactam piperacillin-tazobactam is compared to predefined pharmacokinetic/pharmacodynamic (PK-PD) targets:
  minimum percentage of time during which the free drug concentration remains above the Minimum Inhibitory Concentration (MIC) of the micro-organism should be 50%.
Blood concentrations with maximal antimicrobial activity versus current dosing regimens for ceftazidim | 9/2016 - 12/2021
  Measured concentration of the beta-lactam ceftazidim is compared to predefined pharmacokinetic/pharmacodynamic (PK-PD) targets:
  minimum percentage of time during which the free drug concentration remains above the Minimum Inhibitory Concentration (MIC) of the micro-organism should be 50%.
Pharmacokinetics of vancomycin in patients undergoing intermittent hemodialysis | 9/2016 - 12/2021
  Population pharmacokinetic modeling is performed based on the measured vancomycin concentrations, to end up with a calibrated kinetic model. The model is fitted on the measured vancomycin concentrations in order to determine the model parameters: distribution volume and (inter)dialytic elimination rate constant and clearance.
Pharmacokinetics of teicoplanin in patients undergoing intermittent hemodialysis | 9/2016 - 12/2021
  Population pharmacokinetic modeling is performed based on the measured teicoplanin concentrations, to end up with a calibrated kinetic model. The model is fitted on the measured teicoplanin concentrations in order to determine the model parameters: distribution volume and (inter)dialytic elimination rate constant and clearance.
Pharmacokinetics of amoxicillin-clavulanic acid in patients undergoing intermittent hemodialysis | 9/2016 - 12/2021
  Population pharmacokinetic modeling is performed based on the measured amoxicillin-clavulanic acid concentrations, to end up with a calibrated kinetic model. The model is fitted on the measured amoxicillin-clavulanic acid concentrations in order to determine the model parameters: distribution volume and (inter)dialytic elimination rate constant and clearance.
Pharmacokinetics of piperacillin-tazobactam in patients undergoing intermittent hemodialysis | 9/2016 - 12/2021
  Population pharmacokinetic modeling is performed based on the measured piperacillin-tazobactam concentrations, to end up with a calibrated kinetic model. The model is fitted on the measured piperacillin-tazobactam concentrations in order to determine the model parameters: distribution volume and (inter)dialytic elimination rate constant and clearance.
Pharmacokinetics of ceftazidim in patients undergoing intermittent hemodialysis | 9/2016 - 12/2021
  Population pharmacokinetic modeling is performed based on the measured ceftazidim concentrations, to end up with a calibrated kinetic model. The model is fitted on the measured ceftazidim concentrations in order to determine the model parameters: distribution volume and (inter)dialytic elimination rate constant and clearance.

SECONDARY OUTCOMES:
Dialyser extraction rate of vancomycin | 9/2016 - 12/2021
  From dialyser inlet and outlet samples, the extraction ratio is calculated for vancomycin and entered in the kinetic analysis
Dialyser extraction rate of teicoplanin | 9/2016 - 12/2021
  From dialyser inlet and outlet samples, the extraction ratio is calculated for teicoplanin and entered in the kinetic analysis
Dialyser extraction rate of amoxicillin-clavulanic acid | 9/2016 - 12/2021
  From dialyser inlet and outlet samples, the extraction ratio is calculated for amoxicillin-clavulanic acid and entered in the kinetic analysis
Dialyser extraction rate of piperacillin-tazobactam | 9/2016 - 12/2021
  From dialyser inlet and outlet samples, the extraction ratio is calculated for piperacillin-tazobactam and entered in the kinetic analysis
Dialyser extraction rate of ceftazidim | 9/2016 - 12/2021
  From dialyser inlet and outlet samples, the extraction ratio is calculated for ceftazidim and entered in the kinetic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Biesen, PhD, MD, Study Chair — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No